CLINICAL TRIAL: NCT06258018
Title: A Phase I-II Study of Niraparib Plus Temozolomide "One Week on, One Week Off" in Patients With Recurrent Isocitrate Dehydrogenase (IDH) Wild Type Glioblastoma and IDH Mutant Gliomas.
Brief Title: Niraparib and Temozolomide in Patients Glioblastoma
Acronym: ONC-2022-001
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Armando Santoro, MD (Other)
Collaborators: Istituto Clinico Humanitas (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, Professor, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2022-001
Record Dates: First submitted 2024-01-11; First posted 2024-02-14 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Glioma, Malignant
Keywords: Glioma; Niraparib; Temodal
MeSH Terms: conditions — Glioma | interventions — Temozolomide; niraparib

STUDY DESIGN:
Intervention Model Description: The "3+3 method" will be followed in the safety run-in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Niraparib + Temodal Level 0 (Experimental): Niraparib 100 mg/die + TMZ 75 mg/m2 both given for 7 consecutive days, followed by 7 days OFF, in a cycle of 28 days (starting dose).
  Interventions: Drug: Temodal; Drug: Niraparib
- Niraparib + Temodal Level 1 (Experimental): Niraparib 100 mg/die + TMZ 100 mg/m2 both given for 7 consecutive days, followed by 7 days OFF, in a cycle of 28 days.
  Interventions: Drug: Temodal; Drug: Niraparib
- Niraparib + Temodal Level 2 (Experimental): Niraparib 200 mg/die + TMZ 75 mg/m2 both given for 7 consecutive days, followed by 7 days OFF, in a cycle of 28 days
  Interventions: Drug: Temodal; Drug: Niraparib
- Niraparib + Temodal Level 3 (Experimental): Level 3: Niraparib 200 mg/die + TMZ 100 mg/m2 both given for 7 consecutive days, followed by 7 days OFF, in a cycle of 28 days.
  Interventions: Drug: Temodal; Drug: Niraparib
- Niraparib + Temodal Level -1 (Experimental): Niraparib 100 mg given on alternate days for 7 days, followed by 7 days of OFF + TMZ given 75 mg/m2 for 7 consecutive days, followed by 7 days OFF, in a cycle of 28 days.
  Interventions: Drug: Temodal; Drug: Niraparib
- Niraparib + Temodal Expansion Phase (Experimental): Niraparib RP2D dose given on alternate days for 7 days, followed by 7 days of OFF + TMZ given RP2D for 7 consecutive days, followed by 7 days OFF, in a cycle of 28 days.
  Interventions: Drug: Temodal; Drug: Niraparib

INTERVENTIONS:
Drug: Temodal — given orally for 7 consecutive days, followed by 7 days OFF, in a cycle of 28 days
  Other Names: Temozolomide
Drug: Niraparib — given orally in continous

SUMMARY:
The study evaluates safety, tolerability, pharmacokinetics at recommended phase II dose (RP2D) and preliminary antitumor activity of Niraparib + dd-TMZ "one week on, one week off" in patients affected by recurrent GBM IDH wild-type and recurrent IDH mutant (WHO grade 2-4) gliomas.

The treatment will be administered until progressive disease, unacceptable toxicity, consent withdrawal, lost to follow-up or death.

The entire study is expected to last approximately 40 months.

DETAILED DESCRIPTION:
Diffuse malignant gliomas are the most common central nervous system (CNS) primary tumours in adults, characterized by poor prognosis and few treatment options. In the last 15 years, standard treatment consisting of surgery, adjuvant radiotherapy and temozolomide (TMZ)-based chemotherapy has remained unchanged. New therapeutic approaches are urgently needed.

TMZ is a DNA-methylating chemotherapeutic agent with good CNS penetration. Its mechanism of action is increased by either gene promoter methylation or consumption of the methylguanine-DNA methyltransferase (MGMT), an enzyme repairing chemotherapy-induced genome damages.

Alternative, intensified schedules of TMZ (dose-dense TMZ, dd-TMZ) can give patients an increased total dose of drugs per each cycle, progressively consuming MGMT and overcoming resistance of cancer cells to standard first-line schedule. They are usually used at disease recurrence, with a tolerable safety profile. For example, a clinical study testing the 7 day on / 7 day off schedule showed that MGMT activity in blood mononuclear cells decreased at day 8 and progressively recovered during the week-off. This may limit haematological toxicity.

The inhibition of Poly (ADP-ribose) polymerase (PARP) proteins, normally involved in genomic stability, may rationally improve TMZ efficacy. Switching off PARP molecules can block both base-excision repair (BER) system and Poly-ADP ribose-ylation of MGMT (a key process for its function), leading to an amplification in DNA damages. In the subset of Isocitrate dehydrogenase (IDH) 1/2 mutant gliomas, the enzyme leads to 2-hydroxy-glutarate (2HG) accumulation in cancer cells. This onco-metabolite increases sensitivity to DNA damages by alkylating agents and induces a Breast Cncer gene(BRCA)-ness phenotype indeed. Considering all this, the use of PARP inhibitors seems promising even for these patients.

When compared to other PARP inhibitors, Niraparib has peculiar pharmacokinetics proprieties, such as higher volume of distribution (Vd) and blood-brain barrier (BBB) penetration. These characteristics lead to a progressive drug accumulation in brain and other body tissues with standard daily administration, reaching concentration well over that necessary for PARP inhibition. Overall, Niraparib can represent an ideal candidate to explore for treatment of malignant gliomas and a non-continuous administration may lead to a reduced bone marrow exposure, decreasing haematological toxicity without compromising anticancer activity.

Previous clinical experiences have already explored PARP inhibitors combined to TMZ in solid malignancies, with scarce tolerability mainly due to bone marrow exhaustion. In one small trial, a continuous administration of Niraparib in combination with standard schedule TMZ across several cohorts confirmed high rate of hematologic toxicities and interestingly showed signals of activity in glioblastoma (GBM).

Considering the peculiar pharmacokinetics proprieties of Niraparib and the recovery in MGMT activity described for dd-TMZ, investigator speculate that different schedules and doses of the two drugs (compared to the ones approved in clinical practice) may be explored to improve tolerability preserving the synergistic activity.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Ability to understand and willingness to sign an ethics committee approved written informed consent document (or that of legally authorized representative, if applicable).
3. Patients with diagnosis of recurrent\progressive IDH wild-type GBM (WHO 2021, grade 4). All the GBM histological variants are allowed.
4. Patients with diagnosis of recurrent/progressive IDH mutant gliomas (WHO 2021, grade 2-4). Both astrocytoma and oligodendroglioma may be included.
5. Both MGMT methylated and unmethylated patients are allowed.
6. Unequivocal evidence of tumor progression with at least one target lesion based on MRI scan according to Response Assessment in Neuro-Oncology criteria (RANO) or low-grade gliomas (LGGs) Response Assessment in Neuro-Oncology (RANO) criteria for non-enhancing tumors
7. Patients with IDH wild-type GBM (WHO grade 4) must have received at least the standard front-line therapy defined as below:

   - Surgery (biopsy alone is allowed), concomitant radio-chemotherapy (hypo-fractionated regimens are allowed) and maintenance temozolomide chemotherapy (up to 6 cycles completed).
8. Patients with IDH mutant gliomas (WHO 2021 grade 2-4, both astrocytoma and oligodendroglioma may be included) must have received at least:

   - Surgery (biopsy alone allowed), radiotherapy (hypo-fractionated regimens allowed) and/or one chemotherapy line [temozolomide, Procarbazine (PC) scheme].
9. Enrollment of patients after salvage surgery for recurrent disease is allowed if point number 6 is matched.
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 or Karnofsky performance status of ≥ 70.
11. Life expectancy > 12 weeks.
12. Ability to swallow intact solid oral dosage form (without chewing, crushing, or opening).
13. Normal bone marrow and organ function as defined below:

    Neutrophils ≥ 1500/mm3 Platelets ≥ 150x103/mm3 Hemoglobin ≥ 9.0 g/dL Serum creatinine ≤ 1.5 x the upper limit of normal (ULN) or creatinine clearance (CrCl)≥ 40 mL/min (using the Cockcroft-Gault formula) Aspartate aminotransferase (AST) ≤ 2 x ULN Alanine aminotransferase (ALT) ≤ 2 x ULN Bilirubin≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
14. international normalized ratio (INR) ≤ 1.5 x ULN
15. partial thromboplastin time (PTT) ≤ 1.5 x ULN
16. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    Is not a woman of childbearing potential (WOCBP). or Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), from the Screening Visit through at least 180 days after the last dose of study treatment and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The Investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment (see also Appendix A).

    A WOCBP must have a negative highly sensitive pregnancy test (urine or serum, as required by local regulations) within 72 hours prior to the first dose of study treatment. (The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy).
17. A male participant of reproductive potential is eligible to participate if he agrees to the following starting with the first dose of study treatment through at least 90 days (a spermatogenesis cycle) after the last dose of study treatment:

refrain from donating sperm plus, either: be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent or must agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception, as a condom may break or leak, when having sexual intercourse with a WOCBP who is not currently pregnant

Exclusion Criteria:

1. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive the planned therapy (including brain surgery), or interfere with the interpretation of study results.
2. Anticancer treatment within the last 14 days before the start of trial treatment, for example chemotherapy, radiotherapy, immunotherapy. A shorter interval can be approved by the principal investigator, if deemed appropriate.
3. Previous G4 hematological toxicity (anemia, neutropenia, thrombocytopenia) during concomitant and/or adjuvant TMZ treatment.
4. Previous treatment with a PARP inhibitor.
5. Presence of diffuse and unequivocal leptomeningeal or extra-cranial disease.
6. Steroid therapy with dexamethasone > 4 mg daily.
7. Chronic (at least 4 weeks) use of drugs with known risk of QT prolongation.
8. Use of anticoagulant agents at therapeutic dose (e.g. Low-molecular-weight heparin ( LWMH), new anti-coagulation oral drug (NAO) , Warfarin). Prophylactic dose is allowed. Antiplatelet agents are allowed.
9. Known primary immunodeficiency or active HIV.
10. Known active or chronic viral hepatitis indicated by positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus ribonucleic acid (HCV RNA).
11. Clinically significant cardiovascular disease within 6 months prior to enrollment (or randomization), including:

    Prior events including myocardial infarction, pericardial effusion, and myocarditis.

    Prior cardiac arrhythmia including atrial fibrillation and atrial flutter or requiring concurrent use of drugs or biologics with pro-arrhythmic potential.

    New York Heart Association (NYHA) Class II or greater heart failure. If cardiac function assessment is clinically indicated or performed, an Ejection fraction (LVEF) less than normal per institutional guidelines, or < 55%, if threshold for normal is not otherwise specified by institutional guidelines.

    corrected QT interval (QTc) prolongation > 470 millisecond or other significant ECG abnormality noted within 14 days of treatment.

    Uncontrolled hypertension, hypertensive crisis, history of hypertensive encephalopathy or history of posterior reversible encephalopathy syndrome (PRES).

    Clinically significant peripheral vascular disease or vascular disease, including rapidly growing aortic aneurysm or abdominal aortic aneurysm > 5 cm or aortic dissection.

    Unstable angina.
12. Patients with a history of cerebrovascular accident or transient ischemic attack within 6 months prior to study enrollment are not eligible.
13. Evidence of hemorrhage on the baseline MRI or CT scan other than those that are ≤ grade 1 and either post-operative or stable on at least two consecutive scans.
14. Active diverticular disease of active and/or uncontrolled inflammatory bowel disease (IBD).
15. Gastrointestinal disorders that would impact on drug absorption.
16. Prior history of myelodysplastic syndrome (MDS) and/or myeloid acute leukemia (AML).
17. Other invasive malignancy within 2 years prior to entry into the study, except for those treated with surgical therapy only.
18. History of allergy to study drug components or of severe hypersensitivity reactions to any monoclonal antibodies.
19. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
20. Participant is at an increased bleeding risk due to concurrent conditions (e.g., major injuries or major surgery within the past 28 days prior to start of study treatment).
21. Participant has received a live vaccine within 28 days of planned start of study therapy. Coronavirus Disease 19 (COVID19) vaccines that do not contain live viruses are allowed.
22. Participants have received a transfusion (platelets or red blood cells), colony-stimulating factors (e.g., granulocyte macrophage colony-stimulating factor or recombinant erythropoietin) within 4 weeks prior to the first dose of study treatment.
23. Participants must not have had radiotherapy encompassing > 20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
24. Women who are breast-feeding or pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG).
25. Women of childbearing potential not using a medically acceptable means of contraception for the duration of the study and unsterilized males not willing to abide by requirements for contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Escalation Phase : maximum tolerated dose (MTD) | 1 year
  To determine the MTD of the combination of dd-TMZ and Niraparib, established in the first cycle of therapy, in order to determine the recommended phase II dose (RP2D).
Expansion Phase : PFS | 8 months
  To assess the proportion of patients progression-free at 6 months for recurrent IDH wild-type glioblastoma (Cohort 1) and at 8 months for recurrent IDH-mutant lower-grade gliomas (Cohort 2)

SECONDARY OUTCOMES:
pharmacokinetics CMAX | 1 year
  To evaluate the pharmacokinetics proprieties of the combination of dd-TMZ and Niraparib given on a 7d ON/7d OFF schedule at specific time-points during experimental treatment.Niraparib given on a 7d ON/7d OFF schedule
cerebrospinal fluid drug concentration | 1 year
  To evaluate cerebrospinal fluid (CSF) drug concentration of the combination of dd-TMZ and Niraparib given on a 7d ON/7d OFF schedule in those cases where it is safely feasible collecting liquor samples through lumbar puncture and only after patient's appropriate consent.
Adverse event monitoring | 2 years
  To assess the safety and tolerability of the combination of dd-TMZ and Niraparib given at the RP2D on a 7d ON/7d OFF schedule
tumour tissue drug concentration | 2 years
  To evaluate tissue drug concentration schedule and visualized intra-tumor distribution by mass spectrometry imaging in surgical specimen of the combination of dd-TMZ and Niraparib given on a 7d ON/7d OFF from patients who need second surgery after patient's consent.
assess objective response rate (ORR) | 2 years
  To assess objective response rate (ORR) defined as the proportion of patients who achieved partial response or complete response according to RANO criteria and LGGs RANO criteria on a 7d ON/7d OFF schedule
assess disease control rate (DCR) | 2 years
  To assess disease control rate (DCR) defined as the proportion of patients who achieved objective partial response, complete response or stable disease according to RANO criteria and LGGs RANO criteria
assess progression-free survival (PFS) | 2 years
  To assess progression-free survival (PFS) defined as the time from the start of experimental treatment to disease progression according to RANO criteria and LGGs RANO criteria or death from any cause
assess overall survival (OS) | 2 years
  To assess overall survival (OS) defined as the time from start of experimental treatment to death from any cause in patients with recurrent/progressive IDH wild-type glioblastoma (Cohort 1) and IDH mutant lower-grade gliomas (Cohort 2).
magnitude of PFSin cohort 2 | 2 years
  To explore the magnitude of PFS in cohort 2 according to brain MRI features (enhancing vs non-enhancing lesions)
magnitude of ORR in cohort 2 | 2 years
  To explore the magnitude of ORR in cohort 2 according to brain MRI features (enhancing vs non-enhancing lesions)
magnitude of OS in cohort 2 | 2 years
  To explore the magnitude of OS in cohort 2 according to brain MRI features (enhancing vs non-enhancing lesions)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Simonelli, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto clinico humanitas, Rozzano, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamers LM, Stupp R, van den Bent MJ, Al MJ, Gorlia T, Wasserfallen JB, Mittmann N, Jin Seung S, Crott R, Uyl-de Groot CA; EORTC 26981/22981 NCI-C CE3 Intergroup Study. Cost-effectiveness of temozolomide for the treatment of newly diagnosed glioblastoma multiforme: a report from the EORTC 26981/22981 NCI-C CE3 Intergroup Study. Cancer. 2008 Mar 15;112(6):1337-44. doi: 10.1002/cncr.23297. PMID 18213621
- [Background] Weller M, van den Bent M, Preusser M, Le Rhun E, Tonn JC, Minniti G, Bendszus M, Balana C, Chinot O, Dirven L, French P, Hegi ME, Jakola AS, Platten M, Roth P, Ruda R, Short S, Smits M, Taphoorn MJB, von Deimling A, Westphal M, Soffietti R, Reifenberger G, Wick W. EANO guidelines on the diagnosis and treatment of diffuse gliomas of adulthood. Nat Rev Clin Oncol. 2021 Mar;18(3):170-186. doi: 10.1038/s41571-020-00447-z. Epub 2020 Dec 8. PMID 33293629
- [Background] Tan AC, Ashley DM, Lopez GY, Malinzak M, Friedman HS, Khasraw M. Management of glioblastoma: State of the art and future directions. CA Cancer J Clin. 2020 Jul;70(4):299-312. doi: 10.3322/caac.21613. Epub 2020 Jun 1. PMID 32478924
- [Background] Mildenberger I, Bunse L, Ochs K, Platten M. The promises of immunotherapy in gliomas. Curr Opin Neurol. 2017 Dec;30(6):650-658. doi: 10.1097/WCO.0000000000000491. PMID 28984704
- [Background] Nagane M. Dose-dense Temozolomide: Is It Still Promising? Neurol Med Chir (Tokyo). 2015;55 Suppl 1:38-49. PMID 26236801
- [Background] Weller M, Stupp R, Reifenberger G, Brandes AA, van den Bent MJ, Wick W, Hegi ME. MGMT promoter methylation in malignant gliomas: ready for personalized medicine? Nat Rev Neurol. 2010 Jan;6(1):39-51. doi: 10.1038/nrneurol.2009.197. Epub 2009 Dec 8. PMID 19997073
- [Background] Tolcher AW, Gerson SL, Denis L, Geyer C, Hammond LA, Patnaik A, Goetz AD, Schwartz G, Edwards T, Reyderman L, Statkevich P, Cutler DL, Rowinsky EK. Marked inactivation of O6-alkylguanine-DNA alkyltransferase activity with protracted temozolomide schedules. Br J Cancer. 2003 Apr 7;88(7):1004-11. doi: 10.1038/sj.bjc.6600827. PMID 12671695
- [Background] Lal S, Snape TJ. A therapeutic update on PARP inhibitors: implications in the treatment of glioma. Drug Discov Today. 2021 Feb;26(2):532-541. doi: 10.1016/j.drudis.2020.10.029. Epub 2020 Nov 4. PMID 33157194
- [Background] van den Bent MJ, Mellinghoff IK, Bindra RS. Gray Areas in the Gray Matter: IDH1/2 Mutations in Glioma. Am Soc Clin Oncol Educ Book. 2020 Mar;40:1-8. doi: 10.1200/EDBK_280967. PMID 32186930
- [Background] Sulkowski PL, Corso CD, Robinson ND, Scanlon SE, Purshouse KR, Bai H, Liu Y, Sundaram RK, Hegan DC, Fons NR, Breuer GA, Song Y, Mishra-Gorur K, De Feyter HM, de Graaf RA, Surovtseva YV, Kachman M, Halene S, Gunel M, Glazer PM, Bindra RS. 2-Hydroxyglutarate produced by neomorphic IDH mutations suppresses homologous recombination and induces PARP inhibitor sensitivity. Sci Transl Med. 2017 Feb 1;9(375):eaal2463. doi: 10.1126/scitranslmed.aal2463. PMID 28148839
- [Background] Wang P, Wu J, Ma S, Zhang L, Yao J, Hoadley KA, Wilkerson MD, Perou CM, Guan KL, Ye D, Xiong Y. Oncometabolite D-2-Hydroxyglutarate Inhibits ALKBH DNA Repair Enzymes and Sensitizes IDH Mutant Cells to Alkylating Agents. Cell Rep. 2015 Dec 22;13(11):2353-2361. doi: 10.1016/j.celrep.2015.11.029. Epub 2015 Dec 10. PMID 26686626
- [Background] Wang Y, Wild AT, Turcan S, Wu WH, Sigel C, Klimstra DS, Ma X, Gong Y, Holland EC, Huse JT, Chan TA. Targeting therapeutic vulnerabilities with PARP inhibition and radiation in IDH-mutant gliomas and cholangiocarcinomas. Sci Adv. 2020 Apr 22;6(17):eaaz3221. doi: 10.1126/sciadv.aaz3221. eCollection 2020 Apr. PMID 32494639
- [Background] Tateishi K, Higuchi F, Miller JJ, Koerner MVA, Lelic N, Shankar GM, Tanaka S, Fisher DE, Batchelor TT, Iafrate AJ, Wakimoto H, Chi AS, Cahill DP. The Alkylating Chemotherapeutic Temozolomide Induces Metabolic Stress in IDH1-Mutant Cancers and Potentiates NAD+ Depletion-Mediated Cytotoxicity. Cancer Res. 2017 Aug 1;77(15):4102-4115. doi: 10.1158/0008-5472.CAN-16-2263. Epub 2017 Jun 16. PMID 28625978
- [Background] Lu Y, Kwintkiewicz J, Liu Y, Tech K, Frady LN, Su YT, Bautista W, Moon SI, MacDonald J, Ewend MG, Gilbert MR, Yang C, Wu J. Chemosensitivity of IDH1-Mutated Gliomas Due to an Impairment in PARP1-Mediated DNA Repair. Cancer Res. 2017 Apr 1;77(7):1709-1718. doi: 10.1158/0008-5472.CAN-16-2773. Epub 2017 Feb 15. PMID 28202508
- [Background] Hanna C, Kurian KM, Williams K, Watts C, Jackson A, Carruthers R, Strathdee K, Cruickshank G, Dunn L, Erridge S, Godfrey L, Jefferies S, McBain C, Sleigh R, McCormick A, Pittman M, Halford S, Chalmers AJ. Pharmacokinetics, safety, and tolerability of olaparib and temozolomide for recurrent glioblastoma: results of the phase I OPARATIC trial. Neuro Oncol. 2020 Dec 18;22(12):1840-1850. doi: 10.1093/neuonc/noaa104. PMID 32347934
- [Background] Federico SM, Pappo AS, Sahr N, Sykes A, Campagne O, Stewart CF, Clay MR, Bahrami A, McCarville MB, Kaste SC, Santana VM, Helmig S, Gartrell J, Shelat A, Brennan RC, Hawkins D, Godwin K, Bishop MW, Furman WL, Stewart E. A phase I trial of talazoparib and irinotecan with and without temozolomide in children and young adults with recurrent or refractory solid malignancies. Eur J Cancer. 2020 Sep;137:204-213. doi: 10.1016/j.ejca.2020.06.014. Epub 2020 Aug 11. PMID 32795876
- [Background] Sun K, Mikule K, Wang Z, Poon G, Vaidyanathan A, Smith G, Zhang ZY, Hanke J, Ramaswamy S, Wang J. A comparative pharmacokinetic study of PARP inhibitors demonstrates favorable properties for niraparib efficacy in preclinical tumor models. Oncotarget. 2018 Dec 14;9(98):37080-37096. doi: 10.18632/oncotarget.26354. eCollection 2018 Dec 14. PMID 30647846
- [Background] Chugh R, Ballman KV, Helman LJ, Patel S, Whelan JS, Widemann B, Lu Y, Hawkins DS, Mascarenhas L, Glod JW, Ji J, Zhang Y, Reinke D, Strauss SJ. SARC025 arms 1 and 2: A phase 1 study of the poly(ADP-ribose) polymerase inhibitor niraparib with temozolomide or irinotecan in patients with advanced Ewing sarcoma. Cancer. 2021 Apr 15;127(8):1301-1310. doi: 10.1002/cncr.33349. Epub 2020 Dec 8. PMID 33289920
- [Background] Chukwueke UN, Wen PY. Use of the Response Assessment in Neuro-Oncology (RANO) criteria in clinical trials and clinical practice. CNS Oncol. 2019 Mar 1;8(1):CNS28. doi: 10.2217/cns-2018-0007. Epub 2019 Feb 26. No abstract available. PMID 30806082
- [Background] van den Bent MJ, Wefel JS, Schiff D, Taphoorn MJ, Jaeckle K, Junck L, Armstrong T, Choucair A, Waldman AD, Gorlia T, Chamberlain M, Baumert BG, Vogelbaum MA, Macdonald DR, Reardon DA, Wen PY, Chang SM, Jacobs AH. Response assessment in neuro-oncology (a report of the RANO group): assessment of outcome in trials of diffuse low-grade gliomas. Lancet Oncol. 2011 Jun;12(6):583-93. doi: 10.1016/S1470-2045(11)70057-2. Epub 2011 Apr 5. PMID 21474379
- [Background] Rao VU, Reeves DJ, Chugh AR, O'Quinn R, Fradley MG, Raghavendra M, Dent S, Barac A, Lenihan D. Clinical Approach to Cardiovascular Toxicity of Oral Antineoplastic Agents: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Jun 1;77(21):2693-2716. doi: 10.1016/j.jacc.2021.04.009. PMID 34045027
- [Background] van Andel L, Zhang Z, Lu S, Kansra V, Agarwal S, Hughes L, Tibben MM, Gebretensae A, Rosing H, Schellens JHM, Beijnen JH. Liquid chromatography-tandem mass spectrometry assay for the quantification of niraparib and its metabolite M1 in human plasma and urine. J Chromatogr B Analyt Technol Biomed Life Sci. 2017 Jan 1;1040:14-21. doi: 10.1016/j.jchromb.2016.11.020. Epub 2016 Nov 19. PMID 27898364
- [Background] Kim H, Likhari P, Parker D, Statkevich P, Marco A, Lin CC, Nomeir AA. High-performance liquid chromatographic analysis and stability of anti-tumor agent temozolomide in human plasma. J Pharm Biomed Anal. 2001 Jan;24(3):461-8. doi: 10.1016/s0731-7085(00)00466-0. PMID 11199225